CLINICAL TRIAL: NCT03637933
Title: Safety and Efficacy of Endoscopic Tattooing in Colorectal Surgery. India Ink vs Sterile Carbon Particle Suspension. Randomized Clinical Trial.
Brief Title: Endoscopic Tattooing and Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Milone, Principal investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: tattooingunina
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Safety and Efficacy of Tattooing Substance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- India ink tattooing (Active Comparator): Experimental group includes patients undergone to preoperative endoscopic tattooing with Sterile Carbon Particle Suspension.
  Interventions: Procedure: endoscopic tattooing
- Sterile Carbon Particle Suspension tattooing (Experimental): Control group includes patients undergone to preoperative endoscopic tattooing with India Ink.
  Interventions: Procedure: endoscopic tattooing

INTERVENTIONS:
Procedure: endoscopic tattooing — The tattoo has to be placed 1 or 2 cm distal to the lesion and tattooing has to be performed in at least 2 of the 4 quadrants of the bowel. A 0.5-1 mL saline bleb has to be raised submucosally and then a similar quantity of India Ink or Sterile Carbon Particle Suspension has to be injectiected into that bleb.

SUMMARY:
Endoscopic tattooing to facilitate colorectal lesions' identification during laparoscopic surgery is a reliable and widely used technique.

India Ink is the standard option for colonic tattoing. Different studies have been reported significant complications, of which the most common is peritonitis, due to ethylene glycol, phenols and animal-derived gelatine contained in the ink. This local inflammatory reaction is the principal reason of the formation of the adhesions detected during the laparoscopy, that make the intervention more difficult. To prevent infection or inflammatory local reaction India ink solution has to be sterilized and diluted, a cumbersome process. In the last years wide diffusion of another endoscopic ink, Sterile Carbon Particle Suspension, has reduced these complications. Sterile Carbon Particle Suspension is a prepackaged, sterile, FDA-approved formulation of pure carbon particle in suspension, that eliminates the need for preinjection preparation.

In an attempt to evaluate safety and efficacy of endoscopic tattooing in colorectal surgery using two different types of ink, a randomized clinical trial has been designed. Two types of endoscopic ink were evaluated: Sterile Carbon Particle Suspension (Experimental group) and India Ink (Control group) and.

ELIGIBILITY:
Inclusion Criteria:

histologically confirmed malignancy planned for an elective, segmental laparoscopic colectomy.

Exclusion Criteria:

emergency surgery open surgery immune depressant disease immune depressant medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | 6 hours after tattooing
  using VAS Scale (from 1 to 10)
Body Temperature | 6 hours after tattooing
Body Temperature | 24 hours after tattooing
White Blood Count | 6 hours after tattooing
White Blood Count | 24 hours after tattooing
C reactive protein | 6 hours after tattooing
C reactive protein | 24 hours after tattooing
Peritoneal adhesions | During operative colectomy
  Intraoperative adhesions, detected during laparoscopy and classified using Zühlke classification ranging from 0 to 4
Visibility of the tattoo | During operative colectomy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Milone M, Vignali A, Manigrasso M, Velotti N, Sarnelli G, Aprea G, De Simone G, Maione F, Gennarelli N, Elmore U, De Palma GD. Sterile carbon particle suspension vs India ink for endoscopic tattooing of colonic lesions: a randomized controlled trial. Tech Coloproctol. 2019 Nov;23(11):1073-1078. doi: 10.1007/s10151-019-02101-y. Epub 2019 Oct 30. PMID 31667693